CLINICAL TRIAL: NCT01678456
Title: Prospective Registration and Independent Assessment of Incidence, Clinical Relevance and Outcome of Serious Adverse Events (SAE) Registered in the German Competence Network on Atrial Fibrillation
Brief Title: Prospective Registration and Assessment of Serious Adverse Events Within the AFNET
Acronym: AFNET A7
Status: Completed | Type: Observational
Sponsor: Atrial Fibrillation Network (Other)
Responsible Party: Sponsor
Other Study IDs: AFNET_A7
Record Dates: First submitted 2005-09-14; First posted 2012-09-05 (Estimated); Last update posted 2020-09-22 (Actual); Status verified 2012-08

CONDITIONS: Atrial Fibrillation; Assessment of Serious Advers Events; Thromboembolic and Bleeding Complications; Complications of Antiarrhythmic Drugs or Invasive Procedures; Assessment by a Critical Event Committee
Keywords: Atrial Fibrillation; Critical Event Committee; Serious adverse events; Thromboembolic complications; Cardiac and noncardiac complications; Bleeding complications; Acute heart failure; Syncope; Resuscitation
MeSH Terms: conditions — Atrial Fibrillation; Syncope

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective registration and independent assessment of SAE associated with atrial fibrillation such as thromboembolic events, and other cardiac and noncardiac complications by a Critical Event Committee.

DETAILED DESCRIPTION:
Atrial fibrillation (AF), the most common sustained rhythm disturbance, is associated with a significantly enhanced mortality and morbidity due to thromboembolic events, and other cardiac and noncardiac complications. Therefore the "Network of Competence on Atrial Fibrillation (AFNET)" supported by the German Ministry for Education and Research (BMBF) was established in order to collect clinical data on patients (pts) with AF (paroxysmal, persistent, permanent) over a study period of 6 years with an expected sample size of 12,000 pts. Incidence, clinical relevance and outcome after SAE is recorded and assessed by a Critical Event Committee (CEC).

The CEC-members (experts in cardiology and neurology) defined as SAE any death with or without relationship to AF, cardio-embolic events (stroke, peripheral arterial embolism), bleeding complications due to antithrombotic therapy, acute heart failure, syncope, resuscitation; additionally, the complication of interventional strategies for AF-treatment and other AF-independent SAEs.

Over a 3-year follow-up period, during 6-monthly and unscheduled visits, the SAEs are systematically documented, blinded and their relationship to AF will be interpreted in detail by the CEC.

ELIGIBILITY:
Inclusion Criteria:

* Atrial fibrillation documented by ECG not older then one year
* Age > 18 years
* Informed consent

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Real-life population Patients with atrial fibrilation documented within the last 12 months before enrollment
Sampling Method: Non-Probability Sample
Enrollment: 13000 (Actual)
Dates: Start 2004-02; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Oeff, Professor, Principal Investigator — SAE-Zentrum Brandenburg/Havel Germany
Locations (1):
- Staedt. Klinikum, Department of Cardiology, Brandenburg, Germany